CLINICAL TRIAL: NCT05849870
Title: Comparing Frailty Care Pathways in Rural Primary Care: a Feasibility Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID 19 caused delays for this project and is unlikely to be revisited.
Sponsor: Aberystwyth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 16470
Record Dates: First submitted 2023-04-28; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2020-07

CONDITIONS: Frailty
Keywords: primary care; rural; intervention
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Intervention Model Description: A feasibility trial employing a cluster randomized control trial design.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: There will be different people assigned to the delivery and the intervention. The effectiveness of this will be established as part of the feasibility evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Comprehensive Geriatric Assessment (CGA) (Active Comparator): Participants in this arm will undertake a Comprehensive Geriatric Assessment, and will be implemented based on Comprehensive Geriatric Assessment Toolkit for Primary Care Practitioners from the British Geriatrics Society. A personalised action plan will be developed and implemented based on the CGA.
  Interventions: Other: Frailty care pathway for older people in a rural primary care setting
- Integrated Care for Older PEople (ICOPE) (Experimental): Participants in this arm will undertake the assessment recommended by the World Health Organisation, and will be implemented by the publicly available app. A personalised action plan will be developed and implemented based on the ICOPE.
  Interventions: Other: Frailty care pathway for older people in a rural primary care setting
- Identification and Management of frailty and sarcopenia (Experimental): Participants in this arm will undertake the assessment recommended by the International Conference on Frailty and Sarcopenia Research Clinical Practice Guidelines for Identification and Management of physical frailty (ICFSR). A personalised action plan will be developed and implemented based on the ICFSR.
  Interventions: Other: Frailty care pathway for older people in a rural primary care setting
- Functional Fitness Battery (FFB) (Experimental): Participants in this arm will undertake a Functional Fitness Battery, comprising physical assessments on the intrinsic capacity, lifestyle and nutritional status
  Interventions: Other: Frailty care pathway for older people in a rural primary care setting
- Usual Care (No Intervention): Participants in this arm will not receive an intervention, but the usual care provided by the primary care provider.

INTERVENTIONS:
Other: Frailty care pathway for older people in a rural primary care setting — This intervention will take place in different primary care providers in a rural environment. Each provider will have one intervention and a no-intervention group, which will be part of the feasibility evaluation. The intervention will comprise a consultation with the participant, based on the different approaches described in the arm descriptions.
  Arms: Comprehensive Geriatric Assessment (CGA); Functional Fitness Battery (FFB); Identification and Management of frailty and sarcopenia; Integrated Care for Older PEople (ICOPE)

SUMMARY:
Primary Care General Practitioners (GPs) are always looking at ways to improve the care of older people and ways to prevent older people from losing their independence. Pro-active provision of support often involves lifestyle advice and is a potentially important aspect of that, as it supports older people before acute care is needed. It's preventative caring, rather than reactive caring. But, implementing pro-active care is hampered by the high current workload of acute care, the uncertainty of 'what works' and whether patients are responsive to pro-active care plans. This project will explore different ways of providing pro-active support to older people who could be at risk of losing their independence and requiring frequent acute care. The benefits of pro-active care are arguably the greatest in these individuals.

DETAILED DESCRIPTION:
This is randomised control trial design with a cluster randomisation, whereby each cluster (a GP surgery) will have a different intervention. As it's a feasibility study, there will only be one cluster per intervention.

Participants will be recruited from 4 local primary care surgeries, and if participants take part, they will have 4 visits, and will be randomly allocation of an intervention arm, or a control arm receiving usual care.

At the start, the participant would have 2 visits of a maximum of 2 hours to the participant's local GP surgery to undergo a variety of tasks and assessments about the participant's well-being, health and physical functioning. That could lead to an 'action plan' that is implemented. The participant will have the 3rd visit after 3 months, and a final (fourth) visit after 12 months. During the 3rd and 4th visit the participant will repeat various tasks and assessments done in visit 1 and 2.

The project comprises different activities in the different GP surgeries. The project compares different approaches that each surgery takes. Generally, each surgery will assess relevant aspects that are associated with 'getting older' and provide support in the coming months. The specific approaches are based on the Comprehensive Geriatric Assessment, the World Health Organisation's recommendation and resources for the Integrated Care of Older People (ICOPE) model, the recommendations from the International Conference of Frailty and Sarcopenia Research (ICFSR) and the Functional Fitness test battery. All of these approaches would lead to an 'personal care plan' developed by the medical student, with actions that are specific to the participant's circumstances.

ELIGIBILITY:
The study focuses on community-dwelling frail older people (≥ 60 years). Each GP surgery will complete the electronic Frailty Index (eFI) to stratify older people based on their level of frailty (non-frail, mildly frail, and frail). Participants will be stratified into four strata,

* participants without complex care needs and with a relatively low frailty level (non-frail);
* participants with some chronic conditions that could put them at risk in the future (mild frailty)
* frail participants at risk of complex care needs (frailty)
* participants with complex care needs (severe frailty).

Inclusion Criteria:

* adults aged 60 years or older
* mild frailty or frailty based on the eFI,
* without severe cognitive impairment diagnoses,
* not currently taking part in other research or in the previous 6 months,
* willing to provide informed consent

Exclusion Criteria:

1. are terminally ill
2. have severe cognitive or psychological impairments,
3. have experienced a severe, disabling stroke within the previous 6 months
4. are unable to communicate in English.
5. are currently taking part in other research project, or was part of research in the previous 6 months.
6. have experienced a heart attack, or unstable angina within the previous 3 months.
7. already receive advice that includes exercise and diet by health professionals and were referred at discharge for condition-specific rehabilitation (e.g. pulmonary rehabilitation, stroke rehabilitation) within the previous 6 months

Ages: 60 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate (feasibility determination) | 6 months
  The recruitment rate reflects the recruitment method and number of eligible patients and general interest to take part.
Drop out rate (feasibility determination) | 12 months
  The drop out rate reflects the number of participants lost to follow up, response rates and adherence/compliance to the intervention.
Frequency of health care use | 12 months
  The number of hospital admissions and GP visits in the preceding 12 months
electronic Frailty Index | 12 months
  This score reflects the number of accumulated deficits

SECONDARY OUTCOMES:
Physical Activity Level | 12 months
  Quantified by the International Physical Activity Questionnaire (IPAQ)
Usual Walking Speed | 12 months
  The average speed of walking at a usual pace over a short distance of several meters
Grip Strength | 12 months
  Maximal strength assessed using a hand held dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Marco Arkesteijn, PhD, Principal Investigator — Aberystwyth University
Locations (1):
- Aberystwyth University, Aberystwyth, Ceredigion, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The project data will be made public via the Open Science Framework. This will include all IPD that underlie results in a publication
Supporting Information: Study Protocol, CSR
Time Frame: By december 2022, final data set will be made available comprising the primary and secondary outcome variables, potential other variables collected as part of the intervention arms.
URL: https://osf.io/exac7/?view_only=078714fc84394ec08617dde4a6910457

REFERENCES:
- [Background] Dent E, Morley JE, Cruz-Jentoft AJ, Woodhouse L, Rodriguez-Manas L, Fried LP, Woo J, Aprahamian I, Sanford A, Lundy J, Landi F, Beilby J, Martin FC, Bauer JM, Ferrucci L, Merchant RA, Dong B, Arai H, Hoogendijk EO, Won CW, Abbatecola A, Cederholm T, Strandberg T, Gutierrez Robledo LM, Flicker L, Bhasin S, Aubertin-Leheudre M, Bischoff-Ferrari HA, Guralnik JM, Muscedere J, Pahor M, Ruiz J, Negm AM, Reginster JY, Waters DL, Vellas B. Physical Frailty: ICFSR International Clinical Practice Guidelines for Identification and Management. J Nutr Health Aging. 2019;23(9):771-787. doi: 10.1007/s12603-019-1273-z. PMID 31641726
- [Background] de Jong LD, Peters A, Hooper J, Chalmers N, Henderson C, Laventure RM, Skelton DA. The Functional Fitness MOT Test Battery for Older Adults: Protocol for a Mixed-Method Feasibility Study. JMIR Res Protoc. 2016 Jun 20;5(2):e108. doi: 10.2196/resprot.5682. PMID 27324114
- See also: The CGA toolkit for primary care, used in one of the intervention arms — https://www.bgs.org.uk/resources/resource-series/comprehensive-geriatric-assessment-toolkit-for-primary-care-practitioners
- See also: The ICOPE app, used in one of the intervention arms — https://play.google.com/store/apps/details?id=com.universaltools.icope&hl=en_GB